CLINICAL TRIAL: NCT01172444
Title: AN INVESTIGATOR-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY TO ESTABLISH THERAPEUTIC EQUIVALENCE OF 1000 mg MESALAMINE RECTAL SUPPOSITORIES AND CANASA® RECTAL SUPPOSITORIES (1000 mg MESALAMINE, USP) IN THE TREATMENT OF MILD TO MODERATE ULCERATIVE PROCTITIS
Brief Title: Clinical Trial With Mesalamine 1g Suppositories
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MESA-ULP3125
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2015-07

CONDITIONS: Proctitis
Keywords: Mild to Moderate Ulcerative Proctitis
MeSH Terms: conditions — Proctitis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Sandoz Mesalamine 1 g Suppository
  Interventions: Drug: Mesalamine
- Reference (Active Comparator): Canasa 1 g Suppository
  Interventions: Drug: Canasa
- Placebo (Placebo Comparator): Sandoz 1 g Placebo Suppository
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine — Supporitory, Once Daily, Per Rectal for 6 Weeks
  Arms: Test
Drug: Canasa — Suppository, Once Daily, Per Rectal for 6 Weeks
  Arms: Reference
Drug: Placebo — Suppository, Once Daily, Per Rectal for 6 Weeks
  Arms: Placebo

SUMMARY:
An Investigator-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Establish Therapeutic Equivalence of 1000 mg Mesalamine Rectal Suppositories and Canasa® Rectal Suppositories (1000 mg Mesalamine, USP) in the Treatment of Mild to Moderate Ulcerative Proctitis will be conducted in 533 patient with a estimated duration of 18months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, male and female, 18 to 65 years of age 2. Active, mild to moderate UP, with disease activity not to exceed 15 cm beyond the anal verge: the upper disease boundary will be confirmed by flexible sigmoidoscopy/colonoscopy performed within 14 days of the Baseline Visit 3. Newly diagnosed or newly relapsed UP, where newly relapsed UP is defined as UP that has relapsed within less than and equal to 6 weeks prior to the Baseline Visit 4. A Disease Activity Index (DAI) score greater than or equal to 4 and less than or equal to 10 at the Baseline Visit; the DAI must include a Physician's Global Assessment (PGA) sub-score of less than or equal to 2, a rectal bleeding sub-score of greater than or equal to 1 and a mucosal appearance sub-score of greater than or equal to 1 5. Histological confirmation of UP with a Histological Disease Activity Score > or equal to 1 for the biopsy taken from the most severe area of disease during the flexible sigmoidoscopy/colonoscopy performed within 14 days of the Baseline Visit 6. For female patients of child-bearing potential, a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit; all female patients will be considered of child-bearing potential unless they are post-menopausal for at least one year or have been surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) 7. Female patients of childbearing potential must be practicing one of the following methods of birth control and must agree to continue with regimen throughout the study: hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of one full cycle (based on the patient's usual menstrual cycle period) before investigational product administration; total abstinence from sexual intercourse (since the last menses before investigational product administration); intrauterine device; double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream); Male patients must also agree to use acceptable methods of birth control with their female partners, and this may include use of a male condom plus spermicide. 8. Ability to give written informed consent 9. Ability and willingness to comply with study requirements, including dosing procedures, diary completion, and study visits

Exclusion Criteria:

1. Known history of allergic reaction or clinically significant intolerance to aspirin or salicylate derivatives (including mesalamine) or non-active ingredients of the investigational product 2. Onset of UP relapse >6 weeks prior to the Baseline Visit for patients experiencing a relapse of their UP (i.e., patients who are not newly diagnosed) 3. Severe UP as defined by a DAI score of greater than or equal to 11 or a PGA sub-score of 3 4. Histological Disease Activity Score > or equal to 1 for the biopsy taken from the normal tissue above the disease margin during the flexible sigmoidoscopy/colonoscopy performed within 14 days of the Baseline Visit 5. UP with disease involvement greater than 15 cm beyond the anal verge as confirmed on flexible sigmoidoscopy/colonoscopy 6. Prior unsuccessful treatment of active UP or active ulcerative colitis with rectally administered mesalamine preparations of any strength 7. Any prior treatment of UP or ulcerative colitis with any oral 5-aminosalicylic acid product if used at >2 g/day, regardless of treatment outcome 8. Use of local, rectally administered therapies for UP or ulcerative colitis (e.g., suppositories or enemas containing mesalamine, etc.) within 30 days of the Baseline Visit 9. Use of any of the following medications: - Biological therapies (e.g., infliximab) within 90 days of the Baseline Visit - Immunosuppressive/immunomodulating (e.g., azathioprine) medications within 90 days of the Baseline Visit - Oral, intravenous, intramuscular, or rectally administered corticosteroids within 30 days of the Baseline Visit; the use of intranasal and/or inhaled corticosteroids is permitted - Oral 5-aminosalicylic acid products within 7 days of the Baseline Visit, if used at & less than or equal to 2 g/day - Oral, intravenous, or intramuscular antibiotics within 7 days of the Baseline Visit - Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within 7 days of the Baseline Visit; low-dose aspirin (less than or equal to 325 mg/day) taken for cardio-protective reasons is permitted - Antidiarrheals, antispasmodics, and iron therapy within 7 days of the Baseline Visit - Transdermal nicotine products within 7 days of the Baseline Visit 10. A change in regimen (i.e., dosage or frequency of use) of permitted medications within 30 days of the Baseline Visit, or any plans to change the regimen during the course of this study 11. Use or treatment with an investigational drug, therapy, or device within 30 days of the Baseline Visit 12. A planned change in tobacco usage (e.g., smoking, oral tobacco) during the study 13. Female patients who are pregnant, planning a pregnancy, or who are breastfeeding 14. Diseases interfering with the DAI assessment, including but not limited to, hemorrhoids and anal fissures 15. History of Crohn Disease, short bowel syndrome, or bowel surgery (except appendectomy), or active peptic ulcer 16. A positive stool culture for enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, Vibrio, E. coli O157/H7), detection of Clostridium difficile toxin through immunoassay, or enteric parasites and their ova (including Giardia, Cryptosporidium, and Entamoeba histolytica) on routine microscopy at the Screening Visit 17. Significant impairment of renal or hepatic function, as defined by any of the following: - Creatinine >1.5 x Upper Limit Normal (ULN) - Alanine Amino Transferase (ALT) >2.5 x ULN - Aspartate Amino Transferase (AST) >2.5 x ULN 18. Serologic positivity for the Hepatitis B virus (HBV), the Hepatitis C virus (HCV), the Human Immunodeficiency Virus (HIV), or Treponema pallidum (the causative agent of syphilis) 19. Known history of idiopathic / chronic pancreatitis 20. History of active drug or alcohol abuse within the past year, or physical examination findings indicating the same 21. Current clinically significant urinary tract obstruction 22. History of coagulation disorders, including those requiring treatment with anticoagulant drugs (except for aspirin taken at ≤325 mg/day for cardio-protective reasons 23. Current active malignancy or history of malignancy within the past five years, except for cervical carcinoma in situ, squamous or basal cell carcinoma of the skin that has been surgically removed, or prostate cancer that is being managed by watchful waiting (observation alone) 24. History of pelvic irradiation 25. Any other clinically significant abnormal medical condition that in the Investigators judgment would put the patient at increased risk of illness or injury, would interfere with study participation or would interfere with the evaluation or quality of the data 26. Inability or unwillingness to understand and comply with the requirements of the protocol for any reason, including dosing procedures and visit requirements 27. Previous randomization in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
DAI Score | 6 Weeks
  Mean difference in the DAI score between Baseline and the Final Visit.

SECONDARY OUTCOMES:
DAI Score, Improvement, Remission & Histological Disease Activity Score | 3 and 6 Weeks
  * The mean difference in the DAI score and each of the individual DAI parameters between Baseline, Interim and Final Visits
  * Proportion of patients achieving an "improvement", defined as a ≥3 point improvement in overall DAI score and the proportion of patients achieving a "remission", where "remission" is defined as a DAI score of 0-1 at the Interim and Final Visit.
  * The mean difference in the histological disease activity score between baseline and the Final Visit

CONTACTS AND LOCATIONS:
Locations (38):
- India (38):
  - Kamineni Hospitals, 4-1-1227, King Koti Road, Abids, Hyderabad, Andhra Pradesh
  - Nizam's Instiute of Medical Sciences, Department of Gastroenterology, Hyderabad, Andhra Pradesh
  - Andhra Hospitals, Vijayawada, Andhra Pradesh
  - Nagarjuna Hospitals Limited, Vijayawada, Andhra Pradesh
  - Manikya Institute of Gastroenterology and Hepatology, MVV Chambers,203,204, Visakhapatnam, Andhra Pradesh
  - Institute of Digestive and Liver Diseases, Guwahati, Assam
  - Global Liver & Gastroenterology Centre, E-5/24, Opp Arera Petrol Pump, Arera Colony, Bhopal
  - Indira Gandhi Institute of Medical Sciences, Sheikhpura, Patna, Bihar
  - Department of Gastroenterology, Sheth V. S. General Hospital, Ahmedabad, Gujarat
  - Ratandeep Surgical Hospital & Endoscopy Clinic, Ahmedabad, Gujarat
  - Dr. Bhatnagar's Clinic, Ahmedabad, Gujarat
  - Apollo Hospital International Ltd., Ahmedabad, Gujarat
  - Gastro Care Clinic, Rajkot, Gujarat
  - Gastro Care, Surat, Gujarat
  - Gokula Metropolis Clinical Research Center, M.S.Ramaiah Memorial Hospital, New BEL Road, MSRIT Post, Bangalore, Karnataka
  - PVS Memorial Hospital, Kochi, Kerala
  - Sree Gokulam Medical College and Research Foundation, Thiruvanathapuram, Kerala
  - Gut- N-Hepa Care, Indore, Madhya Pradesh
  - KEM Hospital & Research Centre, Department of Surgery, Pune, Maharashtra
  - Midas Institute of Gastroenterology, Rāmdaspeth, Nagpur
  - Department of Gastroentrology, Postgraduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Dr. Nijhawan's Clinic, Jaipur, Rajasthan
  - Sharma Gastroenterology Centre, Jaipur, Rajasthan
  - Kala Endoscopy & Liver Clinic, Jodhpur, Rajasthan
  - Apollo Speciality Hospitals, Lake View Road, K. K. Nagar, Madurai, Tamil Nadu
  - Ajanta Hospital and IVF Center 765, ABC Complex , Kanpur Road, Alambagh, Lucknow, Uttar Pradesh
  - C.S.M Medical University, Department of Surgical Gastroenterology, New Surgical Block (NSB), Lucknow, Uttar Pradesh
  - Dept. of Gastroenterology, Fortis Hospital, B-22, Sector-62, Noida, Uttar Pradesh
  - Samvedna Hospital, B 27/88G, New Colony, Ravindrapuri, Varanasi
  - Anand Multispeciality Hospitals Pvt Ltd, White house, Opp Rajasthan Hospital,Shahibaug, Ahmedabad
  - Leads Medical Center, First Floor, Ozone Complex, Hyderabad
  - Dept. of Gastroenterology & Hepatology, Deccan College of Medical Sciences,Owaisi Hospital & Research Centre, Hyderabad
  - RAI Speciality Care Centre, Jaipur
  - School of Digestive and Liver Diseases, IPGME&R, Kolkata
  - Gastroenterology and Endoscopy Center, Nagpur
  - Senior Consultant-Gastroenterology and Hepatology, Indraprastha Apollo Hospitals, New Delhi
  - Krishna Institute of Medical Sciences Ltd, Secunderabad
  - Liver Clinic, Surat